CLINICAL TRIAL: NCT01444261
Title: Prevention of Iron Deficiency in Breastfed Infants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: University of Iowa (Other)
Responsible Party: Principal Investigator, Ekhard Ziegler, Professor, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BFe10D
Record Dates: First submitted 2011-09-28; First posted 2011-09-30 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Iron Deficiency; Anemia
Keywords: iron deficiency; anemia
MeSH Terms: conditions — Iron Deficiencies; Anemia | interventions — ferrous sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Active Comparator): Fer-in-Sol drops and iron-fortified cereal
  Interventions: Dietary Supplement: Fer-in-Sol
- Control (Other): No intervention
  Interventions: Other: control

INTERVENTIONS:
Dietary Supplement: Fer-in-Sol — Fer-in-Sol drops providing 7.5 mg iron in 0.3 ml per day given from 84 to 168 d of age and iron-fortified cereal
  Arms: Intervention
Other: control — No dietary supplements
  Arms: Control

SUMMARY:
With early screening and appropriate iron supplementation, iron deficiency in the first year of life can be prevented in breastfed infants.

DETAILED DESCRIPTION:
Infants with low ferritin at 1 month are at high risk of iron deficiency. They will receive iron drops starting at 2 months. All other infants are at low risk of iron deficiency. All infants will receive iron-fortified cereal starting at 4 months of age.

ELIGIBILITY:
Inclusion Criteria:

* Term infants
* gestational age 37-42 weeks
* birth weight > 2500 g
* exclusively breastfed at 28 d of age
* intend to breast feed until 9 mo of age

Exclusion Criteria:

* supplemental formula before 4 mo of age

Ages: 4 Weeks to 9 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 219 (Actual)
Dates: Start 2010-12; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Iron deficiency anemia will be prevented in all infants before 5.5 mo of age | 5.5 mo
  Iron deficiency anemia will be defined as plasma ferritin less than 10 ug/L and hemoglobin less than 105 g/L. The expected outcome is there will be no infants with iron deficiency anemia before 5.5 mo of age.

SECONDARY OUTCOMES:
Determine the number of infants with iron deficiency between 5.5 and 9 mo of age | 9 mo
  Iron deficiency will be determined as plasma ferritin less than 10 ug/L. We will determine the number of infants with iron deficiency between 5.5 and 9 mo of age

CONTACTS AND LOCATIONS:
Overall Officials: Ekhard Ziegler, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States